CLINICAL TRIAL: NCT06449742
Title: A Prospective Observational Study of Artificial Intelligence Morphometric Evaluation of Vertebral Fractures
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Di Filippo, Medical Physician Specialist in Endocrinology, IRCCS San Raffaele
Other Study IDs: SMORFIA
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Vertebral Fracture; Osteoporosis
MeSH Terms: conditions — Spinal Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing to CT abdomen-chest: Patients undergoing to CT abdomen-chest study at the UO of Radiology of the IRCCS San Raffaele Hospital for clinical indications not related to osteo-metabolic pathology.
  Patients will be evaluated for vertebral fractures both through the radiological medical evaluation with automatic 3D reconstruction of the thoracic and lumbar spine and through application of the AI software NanoxAIHealthVCF, NANO-X IMAGING LTD on abdomen-chest CT studies.
  Interventions: Diagnostic Test: AI software and automatic 3D reconstruction

INTERVENTIONS:
Diagnostic Test: AI software and automatic 3D reconstruction — Radiological medical evaluation with automatic 3D reconstruction of the thoracic and lumbar spine and through application of the AI software NanoxAIHealthVCF, NANO-X IMAGING LTD on abdomen-chest CT studies.

SUMMARY:
The study will be conducted as a monocentric observational prospective study design wants to evaluate the prevalence of vertebral fractures in the cohort of patients that perform a chest-abdomen CT for medical indication other than osteometabolic pathologies.

DETAILED DESCRIPTION:
This study aimed to evaluate the prevalence of vertebral fractures in a cohort of patients that perform a chest-abdomen CT for medical indication other than osteometabolic pathologies.It is estimated that 250 patients will be enrolled (Patients will be enrolled in retrospective and prospective way between 01/03/2025 and 28/02/2026. The presence of one or more vertebral fractures will be evaluated through the radiological medical assessment with automatic 3D reconstruction of the thoracic and lumbar spine and by application of the AI software NanoxAIHealthVCF NANO-X IMAGING LTD on abdomen-chest CT studies.

Clinical, anthropometric, and anamnestic data will be collected from patients undergoing CT assessments. These data will be collected on the day of the radiological examination.

There will be only one evaluation at the time of the CT scan. Only in case of fracture detection, via radiological medical assessment and/or via AI software, the patient will be subsequently evaluated in the Endocrinology Unit as for standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects
2. Age ≥ 50 years
3. Clinical and medical history data available at abdomen-chest CT evaluation
4. Signature of informed consent to the study

Exclusion Criteria:

1. Hospitalized patients
2. Patients known to have osteo-metabolic diseases.
3. with primary and/or acquired immunodeficiency states, and/or severe impairment of general clinical condition (e.g. metastatic neoplasms; immunosuppressive therapies; worsening/reacute/compensated chronic diseases; moderate-severe renal failure)
4. Patients unable to understand and sign the Informed Consent.

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Male patients, with an age ≥ 50 years old, that perform CT scan, without osteo-metabolic conditions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of fractures detected with CT scans trough AI software and 3D reconstruction | from 01/03/2025 to 28/02/2026
  The UO of Endocrinology, in collaboration with the UO of Radiology of the IRCCS San Raffaele Hospital, proposes to assess the prevalence of vertebral fractures prospectively in the population afferent to our hospital to perform abdomen-chest CT studies through the radiological medical evaluation with automatic 3D reconstruction of the thoracic and lumbar spine and the application of the AI software cNanoxAIHealthVCF, NANO-X IMAGING LTD.